CLINICAL TRIAL: NCT05033353
Title: The Ventilatory Influence on Cerebral Oxygenation in Patients Undergoing VATS
Brief Title: Ventilatory Influence on Cerebral Oxygenation During VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Mogahed, Associate professor, Tanta University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Ministry of health
Record Dates: First submitted 2021-08-23; First posted 2021-09-02 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Thoracic Diseases
Keywords: OLV
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization was done by sealed envelope method and the patients were divided into two groups; group I (targeted EtCO2 32-38 mmHg) and group II (targeted EtCO2 39-45 mmHg).
  only the anesthetist knows the group of the patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group I (Active Comparator): Mechanical ventilation was adjusted to maintain an EtCO2 of 33-38 mm Hg in group I regional cerebral oxygen monitoring
  Interventions: Diagnostic Test: Monitoring of regional cerebral oxygenation
- Group II (Active Comparator): Mechanical ventilation was adjusted to maintain an EtCO2 of 39-45 mm Hg in group II regional cerebral oxygen monitoring
  Interventions: Diagnostic Test: Monitoring of regional cerebral oxygenation

INTERVENTIONS:
Diagnostic Test: Monitoring of regional cerebral oxygenation — Regional cerebral oxygenation was monitored using near-infrared spectroscopy (O3TM, Masimo, Irvine, CA) placed on the patient's forehead.

SUMMARY:
During (OLV) in (VATS) ; many physiological factors may increase risk of hypoxemia such as positioning and intrapulmonary shunt thus compromising cerebral blood flow and oxygenation, resulting in postoperative neurocognitive dysfunctions. The authors hypothesized that increasing (EtCO2) is the most convenient and powerful method for the management of cerebral desaturation. Methods: Seventy patients undergoing VATS were enrolled in this randomized controlled trial. Mechanical ventilation was adjusted to maintain an EtCO2 of 33-38 mm Hg in group I and an EtCO2 of 39-45 mm Hg in group II. Regional cerebral oxygenation was monitored using near-infrared spectroscopy (O3TM, Masimo, Irvine, CA) placed on the patient's forehead.

DETAILED DESCRIPTION:
All patients were operated on by the same surgical team. Patients with severe bronchial asthma, chronic obstructive pulmonary disease, severe renal insufficiency, severe liver dysfunction, cerebrovascular disease, coagulopathy, uncontrolled diabetes mellitus, uncontrolled hypertension or cardiovascular disease, mental disabilities, hearing impairment were excluded. Patients were seen on the day of surgery in the preoperative area prior to administration of premedication. A 16 or 18-gauge peripheral venous cannula and a 20-gauge radial artery were inserted to all patients preoperatively. Randomization was done by sealed envelope method and the patients were divided into two groups; group I (targeted EtCO2 32-38 mmHg) and group II (targeted EtCO2 39-45 mmHg).

In the operating room, Patients were monitored by 5 lead electrocardiogram, invasive arterial blood pressure (IABP) through the arterial catheter and (Masimo®, Irvine, CA) which provides non-invasive continuous technologies for monitoring and measuring many physiological variables such as arterial oxygen saturation (SpO2), heart rate (HR) and hemoglobin concentration (Hb%) from the (RD Rainbow® SET Pulse Co-Oximeter), end tidal CO2 by capnometer (Nomoline sampling line Masimo ®, CA), noninvasive blood pressure, body temperature, (O3 ®, Masimo, Irvine, CA) attached to the patient to provide continuous monitoring of regional cerebral oxygen saturation (rSO2) of the two hemispheres by a near-infrared spectroscopy sensors connected to regional oximetry system. The sensors were placed bilaterally on patient's forehead after the skin of the forehead had been wiped with an alcohol swab and allowed to dry as recommended by the manufacturer, and (SedLine ®, Masimo, CA) brain function monitoring by Patient State Index (PSI) which is a processed EEG parameter affected by the anesthetic agents.

Before general anesthesia, an epidural catheter was inserted at T5, 6 or T6, 7 interspace and a test dose of 3 ml of 2% lidocaine with epinephrine was given to exclude intrathecal or intravascular positioning of the catheter, for perioperative administration of 4-8 ml/ h of bupivacaine 0.125%. After preoxygenation for 2 minutes, anesthesia was induced in all patients with propofol 1.5-2 mg /kg, fentanyl 3-5 micg/ kg, and rocuronium 0.6-0.8 mg/ kg. A left-sided double-lumen tube (DLT) (39F for males and 37F for females) (Broncho-Cath; Mallinckrodt Medical Ltd, Athlone, Ireland) was used for endotracheal intubation and checked by fibreoptic bronchoscope (Olympus company, Tokyo, Japan) and auscultation. The patient was then positioned in left or right lateral decubitus position according to the surgical side and the DLT was rechecked again. Maintenance anesthesia was provided by sevoflurane to keep a patient state index (Psi) measured by (SedLine, Masimo®, CA) level between 25-50. Additional doses of fentanyl to a total of 7-15 micg/kg and rocuronium boluses were given to control the depth of anesthesia and to maintain stable neuromuscular block.

Initially, all patients were applied with two-lung ventilation using a constant-flow, volume-controlled ventilation mode with a tidal volume 8 mL/kg of the actual body weight, an inspiratory to expiratory (I:E) ratio of 1:2, a respiratory rate of 12 breaths/min, oxygen flow rate of 1.5 L/min, and FiO2 (fraction of inspiratory oxygen) of 1.0 without PEEP. OLV was initiated with skin incision, and the tube lumen of the dependent non ventilated lung was opened to room air. During OLV, tidal volume was reduced to 7 mL/kg, respiratory rate of 12-15 breaths/min, PEEP of 5 cm H2 O, FiO2 of 1.0, oxygen flow rate of 1.5 L/min, I:E 1:2. Then patients were assigned a ventilation strategy designed to achieve an EtCO2 of 32-3 8mm Hg or of 39-45mmHg in group I or II respectively throughout the intraoperative period by (MAQUET FLOW i anesthesia delivery system). This could be achieved by changing the respiratory rate and inspiratory: expiratory (I:E) ratio . rSO2 values obtained and After achieving and maintaining the target EtCO2 for 3 minutes baseline %ΔrSO2 was considerd and recorded every 10 minutes till the end of surgery. Although the data were available to both the anesthetist, there were no specific recommendations made on possible interventions by the study team. Peak inspiratory pressure (PIP) was monitored using a side stream spirometry device (MAQUET FLOW-i). If PIP >30 cmH2O, the volume controlled ventilation mode was changed to a pressure-controlled mode to achieve a targeted VT. Intraoperative fluid replacement by lactated Ringer's solution or hydroxyethyl starch solution was infused at rate of 8-10 ml/kg/h.

rSPO2, PSi, SpO2, mean BP, and HR were recorded before anesthesia, 5 minutes after intubation, 5 minutes after putting the patient in lateral position, after initiating OLV, after achieving and maintaining this target ETCO2 for 3 minutes, and every 10 min till the end of surgery . Hypotension (defined as more than 20% drop in mean ABP from baseline values obtained on admission to the operating room) was treated with ephedrine in 4 mg increments. We used ephedrine rather than phenylephrine as a previous study showed that cerebral oxygen saturation decreases after phenylephrine but remains unaffected after ephedrine in anaesthetized patients.

ABG analysis by (ABL 800, Radiometer, Copenhagen, Denmark. PaO2, PaCO2 , pH, serum lactate, HCO3 concentration, haemoglobin concentration (Hb) ,and sodium and potassium ion concentrations. ABG was performed before anesthesia, after induction of anesthesia when the patient was in supine position, after positioning in the lateral decubitus position during two lung ventilation (TLV), 15 minutes after one lung ventilation (OLV) and every 15 minutes till the end of surgery. All the patients were in lateral position with head down 10º during surgery. If SpO2 decreased below 92% and lasted 30 seconds during OLV, surgery was temporarily interrupted and two-lung ventilation was resumed. At the end of surgery patient turned supine and neuromuscular block was antagonized with sugamadex 2mg/kg. At the time of closure of thoracic cavity, two-lung ventilation was started and both lungs were re-expanded by hand bagging in all patients. Aldrete scores were recorded by post anesthesia care unit (PACU) nurses blinded to group assignment on arrival to the PACU and then every 15 min thereafter until discharge from PACU. Patients were followed up for any complications of lung during their hospital stays. Delirium was assessed using a validated and widely used Confusion Assessment Method (CAM) rating scale, adapted from Inouye et al, immediately on arrival to hospital, then within 18-24 hours after surgery. Diagnosis of delirium requires the presence of both acute onset with fluctuating course and inattention, together with either disorganized thinking or altered level of consciousness. A single trained interviewer, blinded to randomization and proficient and trained in CAM, conducted all the assessments preoperatively when each patient arrived at the hospital and on the next day after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-65 years old
* Patients withASA I and II
* Patients with body mass index (BMI) 21-29 kg/m2
* Patients with admitted for elective VATS requiring OLV for about 1-1.5 h

Exclusion Criteria:

* Patients with severe bronchial asthma
* Patients with chronic obstructive pulmonary disease
* Patients with severe renal insufficiency
* Patients with severe liver dysfunction
* Patients with cerebrovascular disease
* Patients with coagulopathy, uncontrolled diabetes mellitus
* Patients with uncontrolled hypertension
* Patients with cardiovascular disease
* Patients with mental disabilities
* Patients with hearing impairment were excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Effect of changing end tidal CO2 on the regional cerebral oxygen saturation % | 5 months
  Intraoperative ventilatory parameters will be adjusted to attain two different end tidal CO2 and the effect on the regional cerebral oxygen saturation % detected
Heart rate | 5 months
  Intraoperative heart rate (beat per minute) monitoring allover the surgery
Blood pressure | 5 months
  Intraoperative blood pressure (mmHg) monitoring allover the surgery

SECONDARY OUTCOMES:
Postoperative cognitive function | 5 months
  Postoperative cognitive function and monitored by a trained personnel

CONTACTS AND LOCATIONS:
Overall Officials: Mona M Mogahed, Principal Investigator — Tanta University
Locations (1):
- Mona Mohamed Mogahed, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No